CLINICAL TRIAL: NCT06187103
Title: Evaluation of Improved Onboard Patient Imaging With the HyperSight Platform on TrueBeam 4.1
Brief Title: Evaluation of Improved Onboard Patient Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2023-05
Record Dates: First submitted 2023-11-27; First posted 2024-01-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer; Breast Cancer; Upper Gastrointestinal Cancer; Lung Cancer; Pelvic Cancer
Keywords: CBCT
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-site feasibility study designed to generate data describing the quality and applicability of on-couch high-performance CBCT imaging technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HyperSight Imaging arm (Experimental): Subjects are imaged with the new HyperSight CBCT imaging system.
  Interventions: Device: HyperSight Imaging

INTERVENTIONS:
Device: HyperSight Imaging — Patients receive standard of care radiation treatment on a Varian TrueBeam system equipped with HyperSight CBCT imaging. Images acquired for daily patient positioning from two different treatment fractions - typically one near the beginning of the treatment course and one at about the halfway point - will be analyzed for the study.

SUMMARY:
The primary objective of radiation therapy is to deliver a therapeutic dose of radiation precisely to the target while minimizing exposure to healthy surrounding tissues. Image-guided radiation therapy (IGRT) involves acquiring cone beam computed tomography (CBCT) scans just before or during treatment sessions. By comparing the CBCT images with the reference images from the treatment planning process, clinicians can make necessary adjustments to ensure precise targeting and account for any changes that may have occurred since the initial planning. Conventional CBCT technology is, however, limited by several factors including long acquisition times that result in motion artifacts in the image, smaller fields of view that limit the volume of anatomy that can be imaged, poor image quality that limits soft tissue visibility, and artifacts created by dense metal implants. This study will evaluate a novel CBCT imaging solution ("HyperSight") that has the potential to address the challenges of conventional CBCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide written consent.
2. Patient is at least 18 years of age at the time of consent.
3. Patient has biopsy confirmed malignancy and recommendation for definitive or palliative radiation to the head and neck, breast, lungs, upper GI structures, or pelvis.
4. Patient has ECOG performance status 0-2.
5. Patient will be receiving radiation therapy at University of Maryland Medical Center, Department of Radiation Oncology.

Exclusion Criteria:

1. Patient is pregnant or attempting pregnancy.
2. Patient has known genetic pre-disposition for sensitivity to radiation (e.g., Li Fraumeni).
3. Patient receives palliative radiation for 5 or fewer fractions.
4. Patient is part of a vulnerable population (per ISO 14155:2020, "individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response"). This includes prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fraction of patients whose HyperSight CBCT images meet the criteria for CBCT-based treatment planning. | 1 year
  To evaluate the feasibility of HyperSight CBCT as a method for CBCT-based re-planning by measuring the fraction of patients whose HyperSight imaging meets criteria for potential CBCT-based treatment planning using HyperSight CBCT. The criteria include visibility of all key anatomical structures, image quality sufficient to contour anatomical structures, and clinically acceptable dose accuracy.

SECONDARY OUTCOMES:
Fraction of patients whose HyperSight CBCT images meet the criteria for CBCT-based treatment planning by anatomical site | 1 year
  To break down the fraction of patients that meet criteria for potential CBCT-based treatment planning using HyperSight CBCT by anatomical site (head/neck, breast, lungs, upper GI tract, and pelvis).
Image noise | 1 year
  To evaluate the imaging noise in HyperSight CBCT using clinical images and to compare this aspect of image quality to simulation CT images.
Image low-contrast resolution | 1 year
  To evaluate contrast between adjacent anatomical structures in HyperSight CBCT using clinical images and to compare this aspect of image quality to simulation CT images.
Image contrast-to-noise ratio | 1 year
  To measure the contrast-to-noise ratio of HyperSight CBCT using clinical images and to compare this aspect of image quality to simulation CT images.
Qualitative assessment of motion artifacts | 1 year
  To evaluate the severity of motion artifacts observed in HyperSight CBCT using clinical images and to compare motion artifacts to simulation CT. Qualitative assessments will be performed by independent observers using a 5-point Likert scale.
Qualitative assessment of metal artifacts | 1 year
  To evaluate the severity of metal artifacts observed in HyperSight CBCT in head & neck patients with dental fillings and pelvis patients with hip prostheses and compare metal artifacts between HyperSight CBCT and simulation CT. Qualitative assessments will be performed by independent observers using a 5-point Likert scale, with a score of 1 representing very severe metal artifacts and a score of 5 representing little or no artifact..
Comparison of anatomical structure contours defined on HyperSight and conventional imaging. | 1 year
  To evaluate concordance of anatomical structures contoured on HyperSight with anatomical structures contoured on simulation CT as measured by the Dice Similarity Coefficient.
Comparison of anatomical structure contours defined on HyperSight and conventional imaging. | 1 year
  To evaluate concordance of anatomical structures contoured on HyperSight with anatomical structures contoured on simulation CT as measured by Hausdorff Distance.
Breath hold tolerance | 1-9 weeks
  To evaluate the number of breath holds required for patients with breast, thoracic, and upper GI malignancies during HyperSight CBCT imaging.
Patient experience of HyperSight imaging | 1-9 weeks
  To evaluate patient experience of HyperSight imaging. Patients will be asked to fill out a questionnaire. Questions will use a 5-point Likert scale.
Impact of noise suppression | 1 year
  HyperSight CBCT images will be reconstructed with different levels of noise suppression and compared qualitatively to CT simulation images of the same patient to identify regions adversely affected by too much or too little noise suppression. This evaluation will be performed for 1-2 subjects in each anatomical region.
Effectiveness of AI auto-contouring | 1 year
  The ability of AI auto-contouring to accurately contour structures on Hy[erSight CBCT will be evaluated (i) via qualitative user feedback on the accuracy of the auto-generated contours, and (ii) quantitatively using overlap metrics (Hausdorff Distance and Dice Similarity Coefficient) to compare auto-generated critical organs at risk to anatomical structures manually contoured on HyperSight CBCT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No